CLINICAL TRIAL: NCT03469219
Title: Serum Granulysin as a Possible Key Marker to Detect the Severity of Psoriasis
Brief Title: Serum Granulysin Level as a Marker to Detect the Severity of Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin Sayed, Principal Investigator, Assiut University
Other Study IDs: SGLPSS
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Psoriasis Vulgaris
Keywords: granulysin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1. Blood samples will be taken from peripheral veins for all subjects.
  2. Punch tissue biopsy will be taken from lesional and perilesional skin for a number of patients in the study group and normal tissue samples for a number of control group subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: patients with psoriasis vulgaris. measuring serum granulysin level for all patients and tissue granulysin level in lesional and perilesional skin for a number of patients using Enzyme Linked Immunosorbent Assay.
- Control group: Healthy volunteers. measuring serum granulysin level for all healthy volunteers and tissue granulysin level for a number of them using Enzyme Linked Immunosorbent Assay.

SUMMARY:
Psoriasis is a chronic inflammatory and proliferative papulosquamous skin disease of unknown cause,overexpression of Anti Microbial Peptides is characteristic of psoriasis.

Granulysin is a cytolytic and proinflammatory peptide that belongs to a family of saposin-like, lipid binding antimicrobial peptides, and localized in the granular compartments of cytotoxic T lymphocytes and natural killer cells,Patients with psoriasis had high tissue granulysin expression, which increased with increased clinical severity of the disease.

The aim of the study is to measure serum granulysin level and correlate with severity of psoriasis and tissue level of granulysin.

DETAILED DESCRIPTION:
The pathogenesis of psoriasis involves dynamic interactions between multiple cell types and numerous cytokines in response to triggers in genetically predisposed individuals leading to activation of T cells and their migration into skin, in addition to dysregulation of immunological cell function, keratinocyte proliferation takes place.

Psoriatic lesions are densely infiltrated by T cells and dendritic cells , the majority of T cells in the dermis are T-helper cells, while T cytotoxic cells predominate in the epidermis. T helper1 secrets cytokines, such as interferon gamma, tumor necrosis factor-alpha and interleukin 12. Recently discovered population of T helper cells called T helper17 cells which secrets interleukin 17 and interleukin 22 which stimulates epidermal proliferation, while interleukin 17 is responsible for the release of proinflammatory cytokines, antimicrobial peptides and chemokines.

A significant upregulation of perforin-expressing lymphocytes, especially cytotoxic T cells and natural killer cells, has been observed in psoriatic patients at the systemic and local levels. Perforin is a prototype granular cytotoxic mediator that ensures the quick access of pro-apoptotic molecules, such as granzymes and granulysin, into the target cells to induce apoptosis .

Granulysin is well associated with diverse activities of natural killer cells and cytotoxic T cells in physiological and pathological settings and could be a useful serum marker for monitoring host cell mediated immune cytotoxic responses.

Granulysin contributes toward the defense mechanisms against mycobacterial and viral infections as it can kill microbial pathogens through disruption of their membrane integrity, this can explain why infections is extremely rare in psoriatic lesions as psoriasis had high tissue granulysin expression, which increased with increased clinical severity of the disease.

Granulysin was found in the sera of healthy individuals at minimal concentrations.

No previous studies performed to detect the level of serum granulysin in patients with psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically typical psoriatic lesions of different ages and sex.
* Patients with psoriasis vulgaris .
* Different degrees of severity according to Psoriasis Area and Index (PASI) Score

Exclusion Criteria:

* Pregnant and lactating women.
* Patients received systemic medical treatment in the last one month.
* Patients with associated disease reported to increase the release of granulysin whether systemic e.g(infection, cancer, organ transplantation, autoimmune disease) or skin e.g( lichen planus , steven Johnson syndrome, toxic epidermal necrolysis, viral vesicles) and patients with severe immune deficiency treated by cell therapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Dermatology clinic at Assiut University.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
serum granulysin level | 1 hour
  blood samples will be collected and measuring serum granulysin level using Enzyme Linked Immunosorbent Assay

SECONDARY OUTCOMES:
lesional tissue granulysin level | 24 hours
  punch tissue biopsy will be taken from lesions, and homogenized then granulysin level measured using Enzyme Linked Immunosorbent Assay
perilesional tissue granulysin level | 24 hours
  punch tissue biopsy will be taken from perilesional skin, and homogenized then granulysin level measured using Enzyme Linked Immunosorbent Assay

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Diab, assis prof, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elgarhy LH, Shareef MM, Moustafa SM. Granulysin expression increases with increasing clinical severity of psoriasis. Clin Exp Dermatol. 2015 Jun;40(4):361-6. doi: 10.1111/ced.12560. Epub 2015 Feb 2. PMID 25639185
- [Background] Vicic M, Peternel S, Simonic E, Sotosek-Tokmadzic V, Massari D, Brajac I, Kastelan M, Prpic-Massari L. Cytotoxic T lymphocytes as a potential brake of keratinocyte proliferation in psoriasis. Med Hypotheses. 2016 Feb;87:66-8. doi: 10.1016/j.mehy.2015.12.004. Epub 2015 Dec 12. PMID 26826643
- [Background] Massari D, Prpic-Massari L, Kehler T, Kastelan M, Curkovic B, Persic V, Ruzic A, Laskarin G. Analysis of granulysin-mediated cytotoxicity in peripheral blood of patients with psoriatic arthritis. Rheumatol Int. 2012 Sep;32(9):2777-84. doi: 10.1007/s00296-011-2013-9. Epub 2011 Aug 10. PMID 21830153
- [Background] Ogawa E, Sato Y, Minagawa A, Okuyama R. Pathogenesis of psoriasis and development of treatment. J Dermatol. 2018 Mar;45(3):264-272. doi: 10.1111/1346-8138.14139. Epub 2017 Dec 10. PMID 29226422
- [Background] Endsley JJ, Torres AG, Gonzales CM, Kosykh VG, Motin VL, Peterson JW, Estes DM, Klimpel GR. Comparative antimicrobial activity of granulysin against bacterial biothreat agents. Open Microbiol J. 2009 Jun 5;3:92-6. doi: 10.2174/1874285800903010092. PMID 19587798
- [Background] Murphy M, Kerr P, Grant-Kels JM. The histopathologic spectrum of psoriasis. Clin Dermatol. 2007 Nov-Dec;25(6):524-8. doi: 10.1016/j.clindermatol.2007.08.005. PMID 18021888
- [Background] Nair RP, Ding J, Duffin KC, Helms C, Voorhees JJ, Krueger GG, Bowcock AM, Abecasis GR, Elder JT. Psoriasis bench to bedside: genetics meets immunology. Arch Dermatol. 2009 Apr;145(4):462-4. doi: 10.1001/archdermatol.2009.73. No abstract available. PMID 19380669
- [Background] Ogawa K, Takamori Y, Suzuki K, Nagasawa M, Takano S, Kasahara Y, Nakamura Y, Kondo S, Sugamura K, Nakamura M, Nagata K. Granulysin in human serum as a marker of cell-mediated immunity. Eur J Immunol. 2003 Jul;33(7):1925-33. doi: 10.1002/eji.200323977. PMID 12884856
- See also: The Journal of The Egyptian Women's Dermatologic Society :Does the antimicrobial peptide, granulysin, play a role in decreasing the incidence of secondary bacterial infection in psoriasis? — https://journals.lww.com/jewds/Fulltext/2011/01000/Does_the_antimicrobial_peptide,_granulysin,_play_a.10.aspx?trendmd-shared=0